CLINICAL TRIAL: NCT02184026
Title: Exposure, Relaxation, & Rescripting Therapy-Child
Acronym: ERRT-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Principal Investigator, Cameo Borntrager, Assistant Professor of Psychology, University of Montana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRA-778
Record Dates: First submitted 2013-07-23; First posted 2014-07-08 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Post Trauma Nightmares; Traumatic Stress
Keywords: nightmare; PTSD; trauma; children; Children Age 8 to 13
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exposure, Relaxation, & Rescripting Therapy-Child (Experimental): Exposure, Relaxation, & Rescripting Therapy-Child utilizes behavioral and cognitive therapy techniques of exposure therapy and cognitive restructuring.
  Interventions: Behavioral: Exposure, Relaxation, & Rescripting Therapy-Child

INTERVENTIONS:
Behavioral: Exposure, Relaxation, & Rescripting Therapy-Child — Exposure, Relaxation, & Rescripting Therapy (ERRT) will be conducted once a week for five consecutive weeks for approximately two hours per session. Each treatment session focuses on one of the following topics/skills: psycho-education and investment in treatment, psycho-education, Progressive Muscle Relaxation, diaphragmatic breathing, child-friendly exposure to the trauma-nightmare, and rescription.

SUMMARY:
The study implements a trauma-related nightmare treatment for children aged 8 to 13 years. Relevant outcome progress and outcome measures on symptoms, nightmare distress and duration, academic indicators, and sleep quality will be examined.

DETAILED DESCRIPTION:
Untreated trauma-related nightmares and sleep-related disorders are associated with chronic health problems, burdening both the suffering individual and the health-care system. The study implements an innovative, cost-efficient, nightmare treatment for trauma-exposed children. It is one of the first randomized clinical trials with children, adapting an efficacious adult therapy to a 5-session nightmare treatment for 8-13 year-olds. Trauma nightmares are a mechanism in development and maintenance of secondary post-trauma psychopathology, medical problems, and family dysfunction. Therefore, this treatment may prevent long-term secondary health and behavioral problems. It provides a viable health care option to Montanans, lessening long-term financial, medical, and behavioral health expenses. Scientific models currently view PTSD treatment as primary, often leaving nightmares untreated. That approach does not address the pernicious impact of trauma-nightmares in individuals with sub-threshold PTSD or whose nightmares are a primary condition. The theoretical innovation of this therapy can advance the field's understanding of the development of trauma sequelae.

ELIGIBILITY:
Inclusion Criteria:

* children age 8-13 with PTSD Criterion A event as defined by the DSM-IV and nightmares occurring at least once per week over a minimum of one month
* have a parent or legal guardian who is able to participate in treatment assignments at home and be able to read and speak English

Exclusion Criteria:

* adult, no traumatic experience, no nightmares, apparent psychosis, pervasive developmental disorder, or mental retardation, not able to read and speak English

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2012-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Trauma Related Nightmare Survey - Child Version (TRNS-C) Reflecting change in nightmare frequency, severity, and duration | Participants will be assessed immediately after treatment which occurs on average for 5 weeks, and then will be assessed for follow-ups at 3 months & 6 months post treatment.
  The TRNS-C is a 14-item self-report measure that assesses current sleep quality, frequency, severity, and duration of nightmares, as well as cognitions, emotions, and behaviors related to nightmares in children.

SECONDARY OUTCOMES:
University of California at Los Angeles Post-traumatic Stress Disorder Reaction Index for the Diagnostic and Statistical Manual of Mental Disorders-IV (DSM-IV) (UPID) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The UPID screens for trauma exposure and posttraumatic symptoms among youth 7 to 18 years old. It queries types of trauma exposures, assesses for DSM-IV criteria of traumatic exposure and the past-month frequency of PTSD symptoms and two associated features of PTSD in childhood.
Revised Child Anxiety and Depression Scale (RCADS) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The RCADS is a 47-item scale that corresponds to the DSM-IV anxiety disorders and it incorporates a sub scale for major depression. There is a six-factor structure with the following sub scales: Separation Anxiety Disorder, Social Phobia, Generalized Anxiety Disorder, Obsessive-Compulsive Disorder, Panic Disorder, and Major Depressive Disorder.
Nightmare Distress Questionnaire - Modified (NDQ) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The NDQ is a 13-item self-report measure of nightmare related distress. Higher scores are significantly related to interest in therapy for nightmares.
Pittsburgh Sleep Quality Index (PSQI) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The PSQI is a 19-item self-report measure of sleep quality and disturbance. It queries sleep quality and disturbances over the last month. Seven component scores are generated from this measure including: subjective sleep quality, latency, duration, habitual sleep efficiency, sleep problems, use of sleep medications, and daytime dysfunction.
Strength and Difficulties Questionnaire - Child Version (SDQ) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The SDQ is a self-report instrument designed for completion by 11-16 year-olds. Specifically, children respond to 25 attributes (emotional, conduct, hyperactivity, peer relationships, and prosocial behaviors).
Children's Sleep Habits Questionnaire (CSHQ) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The CSHQ is a 33-item parent-report measure of sleep behavior that can be used by parents of school-aged children. A total score is derived from items from 8 sub scales: Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Wakings, Parasomnias, Sleep-Disordered Breathing, and Daytime Sleepiness.
Strengths and Difficulties Questionnaire - Parent Version (SDQ) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The SDQ has two parent versions designed for 4-10 year-olds and 11-16 year-olds. Specifically, parents respond to 25 attributes (emotional, conduct, hyperactivity, peer relationships, and prosocial behavior).
The Parenting Stress Scale (PSS) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The PSS is an 18-item measure that assesses stress related to parenting (e.g., "I am happy in my role as a parent," "Having child(ren) has been a financial burden").
Pittsburgh Sleep Quality Index - Parent self-report (PSQI) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  Similar to the child version, the adult form of the PSQI is a 19-item self-report measure of sleep quality and disturbance. It queries sleep quality and disturbances over the last month. It will serve as an index of secondary gain from treatment by way of parent's improved sleep quality and quantity.
The McMaster Family Assessment Device (FAD) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  The FAD is a 53-item measure that identifies seven dimensions of family functioning: Problem Solving, Communication, Roles, Affective Responses, Affective Involvement, Behavior Control, and General Functioning.
Academic Grade Point Average (GPA) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  GPA will be collected as a measure of academic performance.

OTHER OUTCOMES:
Trail Making Test | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as fast as possible while still maintaining accuracy. It provides information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning.
Wechsler Intelligence Scale for Children (WISC-IV), Letter-Number Sequencing subtest | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A measure of attention, short-term auditory memory, and processing speed.
Wechsler Intelligence Scale for Children (WISC-IV), Digit Span subtest | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A measure of auditory short-term memory, attention, and concentration.
Child Attention Network Task | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A task designed to test attention shifting, alerting, orienting, and executive control networks.
A Developmental NEuroPSYchological Assessment (NEPSY-II), Animal Sorting subtest | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A measure of attention and executive functions.
A Developmental NEuroPSYchological Assessment (NEPSY-II), Auditory Attention & Response Set subtest | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A measure of attention and executive functions.
A Developmental NEuroPSYchological Assessment (NEPSY-II), Clocks subtest | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A measure of attention and executive functions.
Aimsweb Reading Curriculum-Based Measurement (R-CBM) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A measure designed to be a short (one minute) fluency measure used to regularly monitor the development of early literacy and early reading skills. Results can be used to evaluate individual student development.
Aimsweb MAZE Reading Curriculum-Based Measurement (MAZE-CBM) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A supplemental measure to provide a more complete picture of a child's reading skill. Maze is a multiple-choice task that children complete while reading silently. The first sentence of a 150-400 word passage is left intact. Thereafter, every 7th word is replaced with three words inside parenthesis. The child must choose the correct word.
Peabody Picture Vocabulary Test, Fourth Edition (PPVT-4) | 1 wk pre-treatment & 1 wk, 3 mo, 6 mo post-treatment follow-ups
  A standardized assessment that evaluates receptive language, as an index of cognitive ability.

CONTACTS AND LOCATIONS:
Overall Officials: Cameo Borntrager, Ph.D., Principal Investigator — University of Montana
Locations (1):
- University of Montana, Missoula, Montana, United States